CLINICAL TRIAL: NCT05269836
Title: Surgify2021. Use of Surgify Safety Burr in Hard Tissue Cutting, Head and Spine Area.
Brief Title: Use of Surgify Safety Burr in Hard Tissue Cutting, Head and Spine Area
Status: Completed | Type: Observational
Sponsor: Surgify Medical Oy (Industry)
Responsible Party: Principal Investigator, Nuutti Vartiainen, HUS, Töölö Hospital, Surgify Medical Oy
Other Study IDs: Surgify2021
Record Dates: First submitted 2022-01-25; First posted 2022-03-08 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Spine Surgery; Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Device: Surgify Safety Burr — Use of Surgify Safety Burr in hard tissue cutting, head and spine area

SUMMARY:
Purpose of the study: To evaluate whether the SSB is safe, useful, beneficial and effective in drilling, cutting and removal of bone tissue in neurosurgical and spine procedures.

DETAILED DESCRIPTION:
Sponsored observational clinical pilot study with no control group. Aim is to get a maximum of 20 study subjects, who have disease of the spine or head requiring surgery with bone removal and who are willing to participate into this study.

ELIGIBILITY:
Inclusion Criteria:

* Disease of the spine or head requiring surgery with bone removal
* Ability to understand the purpose and risks of the study and to give written informed consent
* Age 18-70 years

Exclusion Criteria:

* Previous surgery on the same area
* Abnormalities of bone tissue
* Vulnerable patient (such as prisoner, retarded person, person in nursing home, patient in emergency situation)
* Allergy or hypersensitivity to medical-grade stainless steel or any of alloying components
* Problems with blood clotting

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any 18 to 70 -year old patient scheduled to back/head operation can be recruited according to other inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-11-17 (Actual)

PRIMARY OUTCOMES:
To evaluate usability of SSB | Duration is from recruitment until end of the time on recovery ward, approximately 1 day to 1 week.
  Using video material from operations, microphone recording of the surgeon commentary during drilling and questionnaires to surgeon.
To evaluate safety of SSB | Duration is from recruitment until end of the time on recovery ward, approximately 1 day to 1 week.
  AE reporting

SECONDARY OUTCOMES:
To evaluate effectiveness of SSB | Duration is from recruitment until end of the time on recovery ward, approximately 1 day to 1 week.
  Using video material from operations, microphone recording of the surgeon commentary during drilling
To evaluate beneficiality of SSB | Duration is from recruitment until end of the time on recovery ward, approximately 1 day to 1 week
  Questionnaires to surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Nuutti Vartiainen, MD, PhD, Principal Investigator — HUS
Locations (1):
- HUS,Töölö hospital, Helsinki, Finland